CLINICAL TRIAL: NCT03811041
Title: Adolescent Depression Associated With Parental Depression : Screening, Prevalence and Secondary Prevention From the Meeting of Depressed Parents on Primary Care
Brief Title: Adolescent Depression Associated With Parental Depression
Acronym: AdoDesP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The decision was made not to extend the inclusions due to the low inclusion rate since the beginning of the study. The last inclusion took place on 06/22/2020.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC18.0221
Record Dates: First submitted 2019-01-15; First posted 2019-01-22 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PC articulated with MDA (Experimental): Depressed parent encountered in PC for confirmation of depression with Hopkins Symptom Checklist-25 (HSCL25) scale. If confirmed, the adolescent will also be encountered by the GP for a screening test of depression (Adolescent Depression Rating Scale - ADRS). If negative, the patient will go out of the study. If positive, 2 others tests will be performed to study the intensity of the depression (Child depressionInventory - CDI) and the quality of life (Pediatric Quality of Life InventoryTM).Finally, the patient will be oriented to the MDA of Brest and will meet again the GP at 6 and 12 month to answers the same tests.
  Interventions: Other: MDA
- Routine cares (Active Comparator): Depressed parent encountered in PC for confirmation of depression with Hopkins Symptom Checklist-25 (HSCL25) scale. If confirmed, the adolescent will also be encountered by the GP for a screening test of depression (Adolescent Depression Rating Scale - ADRS). If negative, the patient will go out of the study. If positive, 2 others tests will be performed to study the intensity of the depression (Child depressionInventory - CDI) and the quality of life (Pediatric Quality of Life InventoryTM). Finally, the patient will be oriented to the routine cares and will meet again the GP at 6 and 12 month to answers the same tests.
  Interventions: Other: Routine Cares
- Parental depression (Experimental): Parental depression will be studied. Depressed adolescent encountered in MDA of Marseille for confirmation of depression with 3 tests : ADRS, CDI and PedsQL. If positive, the parent will come to the MDA for a screening test of depression (HSCL25). Parents and adolescent are seen only once.
  Interventions: Other: Parental depression

INTERVENTIONS:
Other: MDA — Depressed adolescents of depressed parents will be oriented to the MDA of Brest for depression cares.
  Arms: PC articulated with MDA
Other: Routine Cares — Depressed adolescents of depressed parents will be oriented to routine cares for depression cares.
  Arms: Routine cares
Other: Parental depression — Parents of depressed adolescents will be met for a screening test of depression.
  Arms: Parental depression

SUMMARY:
Depression is difficult to identify, prevent and treat in adolescents because of complex and stigmatized multiform symptoms and pathways of care.

In children the existence of a parental depression is a significant and recognized risk factor for the development of a depression. It is regularly reported that 30% of adolescents of depressed parents have depression themselves. General Practitioners (GP) have significant access to the depression of adults, potentially parents of teenagers. In fact, 20% of patients in the regular active file of one GP have depression. The primary health care system could provide indirect but voluminous and unprecedented access to the identification of adolescent depression at an early stage from the encounter of depressed parents.

The difficulties of articulation between primary care (PC) and mental health devices are demonstrated. They disrupt the care pathways of adolescents detected in PC, prevention, and may even disturb early detection of depression. An organized joint between the PC and a specialized mental health service for adolescents ("Maison Des Adolescents" MDA) could promote the process of screening and preventing depression of adolescents of depressed parents encountered in PC.

In addition, if the effects of parental depression on adolescents are established, they remain complex and interactive. They vary by age and sex of the child but also the sex of the parent. A concomitant study of adolescent and parent depression will provide data to analyze the prevalence of depressed parent adolescent depression and to define risk or protection factors.

AdoDesP study is a cluster randomised trial (randomisation of the GPs) which compare a group of adolescent with PC articulated with mental health service (MDA) and an other group without articulation (routine cares).

A third group of depressed adolescents will be constituted to analyse parental depression of depressed adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Parents of groups 1 and 2 :

  * Major patient consulting his GP
  * Depressed patient
  * Parent of adolescent aged between 11 and 18 years old
* Adolescents of groups 1 and 2 :

  * Aged more than 11 and less than 18 years old
  * Parent included in the study
* Parents of group 3 :

  * Parent of depressed adolescent under care at the MDA of Marseille, included in the study and whose depression is confirmed by HSCL25 scale
* Adolescents of group 3 :

  * Aged more than 11 and less than 18 years old
  * Depressed patient
  * Under care at the MDA of Marseille since less than 1 month

Exclusion Criteria:

* Parents of groups 1, 2 and 3 :

  * Minor patient
  * Enable to give his consent
  * Patient with guardianship or curatorship
  * Non consenting patient
  * Pregnant or nursing mother
* Adolescents of groups 1 and 2 :

  * Aged < 11 or ≥18
  * Parent whose depression isn't confirmed by HSCL25 scale
  * Non consenting adolescent
  * Pregnant or nursing mother
* Adolescent of group 3 :

  * Aged < 11 or ≥18
  * Non depressed adolescent
  * Non consenting patient
  * Pregnant or nursing mother

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Changes in adolescents' depression intensity | Day 0 and Month12
  The depression intensity will be evaluated by Adolescent Depression Rating Scale (ADRS) at Day 0 and Month 12. The investigators will compare its evolution between group 1 (PC articulated with MDA) and 2 (Routine cares).
  Adolescent depression rating scale (ADRS) assesses depression in adolescents in 10 items. The items measure insomnia, anxiety, sadness and fatigability. If ADRS score is less than 4 : low risk of depression, between 4 and 8 : moderate risk of depression and more than 8 : significant risk of depression.

SECONDARY OUTCOMES:
Diagnosis of depression rate | Day 0
  With group 1 and 2, screening rates for depression in adolescents will be evaluated at Day 0
Changes in adolescents' quality of live | Day 0, Month6 and Month12
  The quality of live will be evaluated by Pediatric Quality of Life InventoryTM (PedsQL) scale at Day 0, Months 6 and 12 and the investigators will compare its evolution between group 1 and 2. 3 scores will be calculated : psychosocial health summary score (average score of 15 items), physical health summary score (average score of 8 items) and the total score (average score of all items). Scores are between 0 and 100% and the higher scores indicate better Health-Related Quality of Life.
Prevalence of adolescent depression with depressed parent | Day 0
  With group 1 and 2, the investigators will calculate de prevalence of adolescent depression when a parent is depressed. Adolescent depression will be assessed by Adolescent Depression Rating Scale (ADRS). This scale is composed of 8 true (1)/false(0) questions. The score is the sum of all item. An adolescent is consider depressed when his score is higher than 4.
Prevalence of parental depression with depressed adolescent | Day 0
  With group 3, the investigators will calculate de prevalence of parental depression when a adolescent is depressed. Parental depression will be assessed by Hopkins Symptom Checklist (HSCL25). This scale is composed of 25 questions with 4 answers (1-4). The score is the average score of the 25 items. The parent is considered depressed when the score is higher or equal to 1.75.
Risk and protection factors | Day 0
  With the 3 groups, the investigators will isolate risk and protection factors for adolescent of depressed parents and for parents of depressed adolescents. Sociodemographics informations will be used and protective or risk factors may be highlighted from the study of some of the medico-psychological and social characteristics of families.

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Dr Phan, Brest
  - Dr Volant-Le-Berre, Brest
  - Dr Wauters, Brest
  - Dr AUGUSTIN, Guilers
  - Dr Le Grignou, Guissény
  - Dr Ac'h, Landerneau
  - Dr PITMAN, Landivisiau
  - Dr CHIRON, Le Relecq-Kerhuon
  - Dr CONNAN, Le Relecq-Kerhuon
  - Dr Cazuguel, Locmaria-Plouzané
  - Dr Coat-Gourio, Plougastel-Daoulas
  - Dr NABBE, Plounéour-Trez

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 3 years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement